CLINICAL TRIAL: NCT02864381
Title: A Phase 2, Open-Label, Randomized Study to Evaluate the Efficacy and Safety of GS-5745 Combined With Nivolumab Versus Nivolumab Alone in Subjects With Unresectable or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Study to Evaluate the Efficacy and Safety of Andecaliximab Combined With Nivolumab Versus Nivolumab Alone in Adults With Unresectable or Recurrent Gastric or Gastroesophageal Junction Adenocarcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-296-2013; 2016-001402-41 (EudraCT Number)
Record Dates: First submitted 2016-08-10; First posted 2016-08-12 (Estimated); Results first posted 2020-09-18 (Actual); Last update posted 2020-09-18 (Actual); Status verified 2020-09

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — andecaliximab; Nivolumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Andecaliximab + Nivolumab (Experimental): Andecaliximab 800 mg plus nivolumab 3 mg/kg administered every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent (up to 34 weeks at the time of the primary efficacy analysis; up to 101 weeks at the time of the safety follow-up analysis).
  Interventions: Drug: Andecaliximab; Drug: Nivolumab
- Nivolumab (Active Comparator): Nivolumab 3 mg/kg administered every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent (up to 41 weeks at the time of the primary efficacy analysis; up to 97 weeks at the time of the safety follow-up analysis).
  Interventions: Drug: Nivolumab

INTERVENTIONS:
Drug: Andecaliximab — 800 mg administered via IV infusion
  Other Names: GS-5745
  Arms: Andecaliximab + Nivolumab
Drug: Nivolumab — 3 mg/kg administered via IV infusion

SUMMARY:
The primary objective of this study is to evaluate and compare the efficacy of andecaliximab (GS-5745) in combination with nivolumab versus nivolumab alone in adults with recurrent gastric or gastroesophageal junction (GEJ) adenocarcinoma.

ELIGIBILITY:
Key Inclusion Criteria:

* Histologically confirmed inoperable locally advanced or metastatic adenocarcinoma of the stomach or GEJ which have progressed on at least 1 prior systemic therapy or line of treatment for unresectable/metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance score of ≤ 1
* Measurable disease according to Response Criteria in Solid Tumors (RECIST) v1.1
* Tumor sites that can be accessed for repeat biopsies
* Archival tumor tissue, preferably obtained from the most recent available biopsy; there must be adequate tissue for a Cochran-Mantel Haenszel (CMH) test stratified by programmed death ligand 1 (PD-L1) stratification test, as assessed by central pathologist
* Individuals not receiving anticoagulant medication must have an international normalized ratio (INR) ≤ 1.5 and activated partial thromboplastin (aPTT) ≤ 1.5 x upper limit of normal (ULN)
* Required baseline laboratory data as outlined in protocol

Key Exclusion Criteria:

* Individuals who have received only neoadjuvant or adjuvant therapy for gastric adenocarcinoma
* Radiotherapy within 28 days of randomization
* Uncontrolled intercurrent illness as outlined in protocol
* History of a concurrent or second malignancy except for those outlined in protocol
* Major surgery, within 28 days of first dose of study drug
* Known positive status for human immunodeficiency virus (HIV)
* Known acute or chronic-active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Chronic daily treatment with oral corticosteroids (dose of > 10 mg/day prednisone equivalent) or other immunosuppressive medications within 14 days of randomization
* Known or suspected central nervous system metastases
* Documented myocardial infarction or unstable/uncontrolled cardiac disease within 6 months of randomization
* Serious systemic fungal, bacterial, viral, or other infection that is not controlled or requires intravenous antibiotics
* Current or history of pneumonitis or interstitial lung disease
* Active known or suspected autoimmune disease with exceptions noted in protocol.
* History of bone marrow, stem cell, or allogenic organ transplantation

NOTE: Other protocol defined Inclusion/ Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-09-01 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2019-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (33):
- United States (6):
  - Los Angeles, California
  - San Francisco, California
  - Chicago, Illinois
  - Fort Wayne, Indiana
  - St Louis, Missouri
  - New York, New York
- Australia (4):
  - Albury, New South Wales
  - Wahroonga, New South Wales
  - Douglas, Queensland
  - Hobart, Tasmania
- Belgium (3):
  - La Louvière, Hainaut
  - Ghent, Oost-Vlaanderen
  - Leuven, Vlaams Brabant
- France (3):
  - Brest, Finistère
  - Reims, Marne
  - Villejuif, Val-de-Marne
- Hungary (2):
  - Budapest
  - Debrecen
- Italy (4):
  - Meldola, Forli-Cesena
  - Genova, Ligura
  - Milan, Lombardy
  - Pisa, Tuscany
- Poland (3):
  - Brzozów, Podkarpackie Voivodeship
  - Poznan
  - Warsaw
- Spain (3):
  - Barcelona, Barcelona
  - Majadahonda, Madrid
  - Barcelona
- United Kingdom (5):
  - Bristol
  - Edgbaston
  - London
  - Manchester
  - Sutton

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Shah MA, Cunningham D, Metges JP, Van Cutsem E, Wainberg Z, Elboudwarej E, Lin KW, Turner S, Zavodovskaya M, Inzunza D, Liu J, Patterson SD, Zhou J, He J, Thai D, Bhargava P, Brachmann CB, Cantenacci DVT. Randomized, open-label, phase 2 study of andecaliximab plus nivolumab versus nivolumab alone in advanced gastric cancer identifies biomarkers associated with survival. J Immunother Cancer. 2021 Dec;9(12):e003580. doi: 10.1136/jitc-2021-003580. PMID 34893523

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, and the United States. The first participant was screened on 01 September 2016. The last study visit occurred on 23 August 2019.
Pre-assignment Details: 187 participants were screened.
Groups:
- Andecaliximab + Nivolumab: Andecaliximab 800 mg administered via intravenous (IV) infusion plus nivolumab 3 mg/kg administered via IV infusion every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent (up to 34 weeks at the time of the primary efficacy analysis; up to 101 weeks at the time of the safety follow-up analysis).
- Nivolumab: Nivolumab 3 mg/kg administered via IV infusion every 2 weeks until disease progression, unacceptable toxicity, or withdrawal of consent (up to 41 weeks at the time of the primary efficacy analysis; up to 97 weeks at the time of the safety follow-up analysis).
Period: Overall Study
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Started | 72 | 72
Completed | 0 | 0
Not Completed | 72 | 72
Not completed — Death | 58 | 61
Not completed — Withdrew Consent | 5 | 6
Not completed — Reason Unknown | 7 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Investigator's Discretion | 1 | 0
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Population: The Intent-to-treat Analysis Set included all participants who were randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Andecaliximab + Nivolumab | Nivolumab | Total
Number analyzed (Participants) | 72 | 72 | 144
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (12.1) | 59 (11.8) | 59 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 22 | 45
  Male | 49 | 50 | 99
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted=local regulators did not allow collection of race information.
  Participants
    Race: Asian | 1 | 1 | 2
    Race: Black | 2 | 0 | 2
    Race: White | 55 | 61 | 116
    Race: Not Permitted | 12 | 8 | 20
    Race: Other | 2 | 2 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted=local regulators did not allow collection of ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 2 | 3 | 5
    Ethnicity: Not Hispanic or Latino | 59 | 61 | 120
    Ethnicity: Not Permitted | 11 | 8 | 19
Region of Enrollment [Number; unit: participants]
  United Kingdom | 17 | 18 | 35
  United States | 14 | 14 | 28
  Belgium | 5 | 10 | 15
  France | 9 | 6 | 15
  Poland | 5 | 9 | 14
  Spain | 10 | 4 | 14
  Italy | 8 | 5 | 13
  Australia | 2 | 5 | 7
  Hungary | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants with confirmed overall best response of complete response (CR) or partial response (PR) after starting study drug but before starting any new chemotherapy or radiotherapy as assessed by the investigator according to Response Criteria in Solid Tumors (RECIST) version 1.1. CR was defined as the disappearance of all target lesions and disappearance of all non-target lesions and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 41 weeks
Population: The Intent-to-treat Analysis Set included all participants who were randomized in the study.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 72 | 72
percentage of participants | 9.7 [4.0 to 19.0] | 6.9 [2.3 to 15.5]
Statistical Analysis 1: Comparison: Andecaliximab + Nivolumab vs Nivolumab; Test type: Superiority; p = 0.8, Cochran-Mantel-Haenszel — P-value is derived from Cochran-Mantel Haenszel (CMH) test stratified by programmed death ligand 1 (PD-L1) stratification factor status; Odds Ratio (OR) = 1.5, 95% CI 2-sided [0.4 to 6.1] — Odds Ratio is derived from CMH test stratified by PD-L1 stratification factor status, the Nivolumab alone arm serves as the reference

2. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as the interval in months from the date of randomization to the earlier of the first documentation of definitive disease progression or death from any cause. The first definitive progressive disease (PD) was defined as the first radiation therapy, the first clinical PD, and the first confirmed imaging PD, whichever came first. Participants without PD or death and participants with PD after starting new anti-cancer therapy are censored at the last tumor assessment date.
Time Frame: Andecaliximab + Nivolumab median follow-up time: 7.0 months; Nivolumab median follow-up time: 7.1 months
Population: Participants in the Intent-to-treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 72 | 72
months | 1.840 [1.807 to 2.004] | 1.856 [1.741 to 1.906]
Statistical Analysis 1: Comparison: Andecaliximab + Nivolumab vs Nivolumab; Test type: Superiority; p = 0.306, Log Rank — P-value is derived from log-rank test stratified by PD-L1 stratification factor status; Hazard Ratio (HR) = 0.836, 95% CI 2-sided [0.589 to 1.189] — Hazard ratio is derived from Cox model stratified by PD-L1 stratification factor status, the Nivolumab alone arm serves as the reference

3. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the interval from the date of randomization to death from any cause. Surviving participants are censored at the last date known alive.
Time Frame: Andecaliximab + Nivolumab median follow-up time: 7.0 months; Nivolumab median follow-up time: 7.0 months
Population: Participants in the Intent-to-treat Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 72 | 72
months | 7.162 [4.797 to NA] — Upper 95% Confidence Interval was not reached due to the low number of participants with events. | 5.881 [3.483 to 10.908]
Statistical Analysis 1: Comparison: Andecaliximab + Nivolumab vs Nivolumab; Test type: Superiority; p = 0.312, Log Rank — P-value is derived from log-rank test stratified by PD-L1 stratification factor status; Hazard Ratio (HR) = 0.786, 95% CI 2-sided [0.491 to 1.257] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Duration of Response (DOR)
Description: DOR was defined as the interval from the date of the first response (complete or partial response) was achieved to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: Andecaliximab + Nivolumab median follow-up time: 7.0 months; Nivolumab median follow-up time: 7.1 months
Population: Participants in the Intent-to-treat Analysis Set who achieved CR or PR were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 7 | 5
months | NA [1.807 to NA] — Median and Upper Limit of Confidence Interval (CI) were not estimable due to the low number of participants with events. | NA [2.037 to NA] — Median and Upper Limit of CI were not estimable due to the low number of participants with events.

5. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participants administered a medicinal product, which does not necessarily have a causal relationship with the treatment. TEAEs are events that are defined as AEs with onset dates on or after the first dose of andecaliximab/nivolumab and up to 30 days after permanent discontinuation of andecaliximab or 5 months after permanent discontinuation of nivolumab, or led to premature discontinuation of andecaliximab or nivolumab.
Time Frame: Andecaliximab: First dose date up to last dose (maximum: 101 weeks) + 30 days; Nivolumab: First dose date up to last dose (maximum: 101 weeks) + 5 months
Population: The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 71 | 70
percentage of participants | 98.6 | 97.1

6. Secondary Outcome: Percentage of Participants Who Experienced Treatment-emergent Laboratory Abnormalities
Description: Treatment-emergent (Chemistry, Hematology, Coagulation, and Urinalysis) laboratory abnormalities were graded per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 where: 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening. Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any postbaseline time point, up to and including the date of the last dose of andecaliximab plus 30 days or nivolumab plus 5 months. If the relevant baseline laboratory value is missing, any abnormality of at least Grade 1 observed within the time frame specified above will be considered treatment-emergent. Percentage of participants with any postbaseline Grade 1 or higher laboratory abnormality is reported.
Time Frame: as for outcome 5
Population: Participants in the Safety Analysis Set with available data were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
Number analyzed (Participants) | 71 | 70
percentage of participants
  Alanine aminotransferase increased: number analyzed (Participants) | 70 | 70
  Alanine aminotransferase increased | 20.0 | 27.1
  Alkaline phosphatase increased | 45.1 | 40.0
  Aspartate aminotransferase increased: number analyzed (Participants) | 70 | 70
  Aspartate aminotransferase increased | 30.0 | 28.6
  Blood bilirubin increased | 8.5 | 11.4
  Chronic Kidney Disease | 16.9 | 25.7
  Creatinine increased | 1.4 | 7.1
  Hyperglycemia | 22.5 | 18.6
  Hyperkalemia: number analyzed (Participants) | 70 | 70
  Hyperkalemia | 7.1 | 5.7
  Hypermagnesemia | 2.8 | 1.4
  Hypoalbuminemia | 35.2 | 38.6
  Hypoglycemia | 11.3 | 4.3
  Hypokalemia: number analyzed (Participants) | 70 | 70
  Hypokalemia | 10.0 | 11.4
  Hypomagnesemia | 5.6 | 4.3
  Hyponatremia | 28.2 | 40.0
  Hypophosphatemia | 11.3 | 8.6
  Lipase increased | 11.3 | 8.6
  Serum amylase increased | 9.9 | 7.1
  Activated partial thromboplastin time prolonged: number analyzed (Participants) | 39 | 31
  Activated partial thromboplastin time prolonged | 2.6 | 19.4
  International Normalized Ratio (INR) increased: number analyzed (Participants) | 39 | 32
  International Normalized Ratio (INR) increased | 2.6 | 12.5
  Anemia: number analyzed (Participants) | 71 | 69
  Anemia | 53.5 | 56.5
  Lymphocytes, Typical count decreased: number analyzed (Participants) | 71 | 69
  Lymphocytes, Typical count decreased | 35.2 | 27.5
  Lymphocytes, Typical count increased: number analyzed (Participants) | 71 | 69
  Lymphocytes, Typical count increased | 4.2 | 0
  Neutrophil count decreased: number analyzed (Participants) | 71 | 69
  Neutrophil count decreased | 5.6 | 5.8
  Platelet count decreased: number analyzed (Participants) | 71 | 69
  Platelet count decreased | 8.5 | 5.8
  White blood cell decreased: number analyzed (Participants) | 71 | 69
  White blood cell decreased | 9.9 | 7.2
  Proteinuria (Dipstick): number analyzed (Participants) | 68 | 67
  Proteinuria (Dipstick) | 29.4 | 31.3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: Andecaliximab + Nivolumab median follow-up time: 28.2 months; Nivolumab median follow-up time: 28.4 months; Adverse Events: Andecaliximab: First dose date up to last dose (maximum: 101 weeks) + 30 days; Nivolumab: First dose date up to last dose (maximum: 101 weeks) + 5 months
Description: All-Cause Mortality: The Intent-to treat Analysis Set included all participants randomized in the study. Adverse Events:The Safety Analysis Set included all participants who received at least 1 dose of study drug.
Arm/Group | Andecaliximab + Nivolumab | Nivolumab
All-Cause Mortality (participants affected / at risk) | 61/72 | 62/72
Serious Adverse Events (participants affected / at risk) | 42/71 | 38/70
Other Adverse Events (participants affected / at risk) | 66/71 | 62/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab + Nivolumab (N=71) | Nivolumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 5 | 4
Ventricular fibrillation (Cardiac disorders) | 0 | 1
Hypophysitis (Endocrine disorders) | 1 | 0
Retinal disorder (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 3 | 6
Abdominal pain upper (Gastrointestinal disorders) | 1 | 1
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 3 | 2
Colitis (Gastrointestinal disorders) | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 4 | 4
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 1 | 0
Gastric stenosis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 3
Gastrointestinal obstruction (Gastrointestinal disorders) | 0 | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 3 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 4 | 0
Intestinal perforation (Gastrointestinal disorders) | 1 | 0
Large intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 0 | 2
Melaena (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 3 | 2
Obstruction gastric (Gastrointestinal disorders) | 0 | 2
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestinal obstruction (Gastrointestinal disorders) | 3 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 3 | 1
Complication associated with device (General disorders) | 1 | 0
Euthanasia (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 0 | 2
Oedema peripheral (General disorders) | 0 | 1
Pyrexia (General disorders) | 2 | 2
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Device related infection (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 0
Liver abscess (Infections and infestations) | 1 | 0
Lung abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Postoperative wound infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 1
Septic shock (Infections and infestations) | 1 | 3
Subcutaneous abscess (Infections and infestations) | 1 | 0
Subdiaphragmatic abscess (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 0 | 1
Blood bilirubin increased (Investigations) | 1 | 2
Blood creatinine increased (Investigations) | 0 | 1
Blood magnesium decreased (Investigations) | 0 | 1
General physical condition abnormal (Investigations) | 1 | 0
Transaminases increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 0 | 2
Malnutrition (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Hepatic encephalopathy (Nervous system disorders) | 1 | 0
Myasthenia gravis (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Renal failure (Renal and urinary disorders) | 1 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab + Nivolumab (N=71) | Nivolumab (N=70)
Anaemia (Blood and lymphatic system disorders) | 14 | 14
Abdominal distension (Gastrointestinal disorders) | 4 | 2
Abdominal pain (Gastrointestinal disorders) | 11 | 16
Abdominal pain upper (Gastrointestinal disorders) | 11 | 2
Ascites (Gastrointestinal disorders) | 7 | 4
Constipation (Gastrointestinal disorders) | 18 | 18
Diarrhoea (Gastrointestinal disorders) | 14 | 9
Dry mouth (Gastrointestinal disorders) | 2 | 5
Dyspepsia (Gastrointestinal disorders) | 5 | 2
Dysphagia (Gastrointestinal disorders) | 12 | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 2
Nausea (Gastrointestinal disorders) | 27 | 17
Vomiting (Gastrointestinal disorders) | 22 | 18
Asthenia (General disorders) | 21 | 12
Chest pain (General disorders) | 1 | 4
Fatigue (General disorders) | 22 | 25
Oedema peripheral (General disorders) | 6 | 6
Pyrexia (General disorders) | 10 | 4
Nasopharyngitis (Infections and infestations) | 4 | 0
Oral candidiasis (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 7 | 1
Alanine aminotransferase increased (Investigations) | 4 | 4
Aspartate aminotransferase increased (Investigations) | 4 | 4
Weight decreased (Investigations) | 5 | 7
Decreased appetite (Metabolism and nutrition disorders) | 24 | 20
Dehydration (Metabolism and nutrition disorders) | 2 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 4
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 5 | 7
Hypomagnesaemia (Metabolism and nutrition disorders) | 4 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 6
Back pain (Musculoskeletal and connective tissue disorders) | 11 | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 3 | 4
Dizziness (Nervous system disorders) | 6 | 8
Headache (Nervous system disorders) | 6 | 6
Paraesthesia (Nervous system disorders) | 1 | 4
Anxiety (Psychiatric disorders) | 5 | 2
Insomnia (Psychiatric disorders) | 3 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 8
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 6
Hypotension (Vascular disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (3):
  • Study Protocol (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/81/NCT02864381/Prot_000.pdf
  • Statistical Analysis Plan: Final (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/81/NCT02864381/SAP_001.pdf
  • Statistical Analysis Plan: Follow-up Analysis (2019-06-28): https://cdn.clinicaltrials.gov/large-docs/81/NCT02864381/SAP_002.pdf